CLINICAL TRIAL: NCT02961296
Title: Helicobacter Pylori Antibiotic Susceptibility Testing of Korea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Principal Investigator, Hwoon-Yong Jung, Professor, Asan Medical Center
Other Study IDs: AMC 2016-0467
Record Dates: First submitted 2016-10-26; First posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Helicobacter Pylori Infection; Peptic Ulcer; Lymphoma; Gastric Cancer; Gastritis
Keywords: Helicobacter Pylori
MeSH Terms: conditions — Peptic Ulcer; Lymphoma; Stomach Neoplasms; Gastritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Mucosa on the antrum and body of the stomach.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No intervention will be needed.

SUMMARY:
The purpose of this study is to make nationwide registry for antimicrobial resistance of Helicobacter pylori using single method with agar dilution in Korea.

DETAILED DESCRIPTION:
Backgrounds:

The success rate of Helicobacter pylori eradication in Korea is not sufficient in recent days. The main cause of eradication failure is known as antimicrobial resistance and previous studies showed that resistant rates were different according to the regions in Korea. However, until now, there are not enough studies about the nationwide results for antimicrobial resistance and previous reports used various methods for the resistant test.

Theories and Plans:

The nationwide resistant registry of Helicobacter pylori using standardized single method, agar dilution test, can be useful for the development of new eradication methods to make eradication rate higher. Moreover, the higher rate of Helicobacter pylori eradication can reduce the chance of gastric cancer and also can reduce the medical expenses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 to 79 year person who need the examination of Helicobacter pylori infection during upper gastrointestinal endoscopy.
* No history of Helicobacter pylori eradication.
* No history of antibiotics within one month.
* Person who agree on the consent.

Exclusion Criteria:

* History of antibiotics more than 3 days sequentially within one month.
* History of subtotal gastrectomy.
* Person who does not agree on the consent.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects required to the examination of Helicobacter pylori infection is necessary during upper gastrointestinal endoscopy due to peptic ulcer, lymphoma, gastric cancer, gastritis, et al.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The rate of exceeding the resistance criteria in Helicobacter pylori(H. pylori) antibiotic susceptibility test(Agar dilution method) | 6 more days
  The resistance criterion specifies that Clarithromycin is excess of 1.0 μg/mL, Amoxicillin is excess of 0.5 μg/mL, Metronidazole is excess of 8 μg/mL, Tetracycline is excess of 4 μg/mL, Levofloxacin is excess of 1 μg/mL and Ciprofloxacin is excess of 1 μg/mL.
  All of resistance criteria follow a criteria of NCCLS(National Committee for Clinical Laboratory Standards)

SECONDARY OUTCOMES:
The gap of the rate of the antibiotic resistance to H. pylori by regional groups | 6 more days
The success rate of H. pylori strain separation | 6 more days
  Analyze the case of inseparable H. pylori strain and the reason of failure for culture after H. pylori strain separation.

CONTACTS AND LOCATIONS:
Overall Officials: Hwoon-Yong Jung, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Department of Gastroenterology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No